CLINICAL TRIAL: NCT07258758
Title: Diabetes Intervention Involving Person-centred Nutritional Education (DINE) - Exploring the Benefits and Challenges of a Person-centred Education on the Nordic Diet for Adults With Type 1 Diabetes.
Brief Title: Diabetes Intervention Involving Person-centred Nutritional Education
Acronym: DINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Lasarettet i Enköping (Other)
Responsible Party: Principal Investigator, Elisabeth Stoltz Sjöström, Associate Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-04356-01
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Type 1
Keywords: Nutritional education; Person-centred care; Nordic diet; Diabetes intervention; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized parallel group study
Masking Description: As the participants are actively involved in the education intervention, it is not possible to have a blinded trial, however each group will not receive information about the alternative group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred nutritional education (Experimental): The participants in this arm will attend a person-centred intervention involving a pre-assessment focused on creating partnership in care. This is followed by a nutrition education session on the healthy Nordic diet, and a series of follow-up measures.
  Interventions: Behavioral: Dietary intervention
- Short dietary information (No Intervention): The participants in this arm will receive short dietary information (brochure) at the same level as standard care.

INTERVENTIONS:
Behavioral: Dietary intervention — A person-centred education focussed on creating partnerships in care and shared decision-making.
  Arms: Person-centred nutritional education

SUMMARY:
The overall objective for this project is to evaluate the effects of a person-centred education intervention to promote a healthy, sustainable Nordic diet compared with the current practice of providing short dietary information on health outcomes of adults with Type 1 diabetes. The study will measure the intervention's impact on blood glucose levels, blood lipids, blood pressure, and adherence to a sustainable and healthy Nordic diet.

The main question the trial aims to answer is:

Does a person-centred nutritional education have an impact on glucose time in range for adults with Type 1 diabetes, compared with short dietary information?

The participants will:

* Attend either a person-centred nutrition education (intervention) or receive short dietary information (control group).
* Wear their sensor for continuous glucose monitoring (CGM) throughout the trial.
* Visit the clinic for data collection (blood samples and clinical checks) at the start and end of the trial.
* Keep a four-day food diary, fill out a food frequency questionnaire (FFQ) and estimate their food enjoyment at the start and end of the trial.

DETAILED DESCRIPTION:
The Diabetes Intervention Involving Person-centred Nutritional Education (DINE) trial is a single-centre, randomized parallel group study conducted in Sweden. The trial aims to compare a person-centred intervention involving nutritional education with the current practice of providing short dietary information to adults with Type 1 diabetes. The study period is six months and will assess the effectiveness of the intervention in a real-world setting, rather than under controlled conditions. Due to the active involvement of participants, blinding of study personnel or participants is not possible.

To determine the sample size, a power calculation was performed using the primary endpoint, 'blood glucose time in range' (TIR). The calculation is based on a clinically relevant change in TIR (8%) from intervention to the six-month follow-up. The proposed enrolment is 54 participants to achieve sufficient power (80%) to test the primary hypothesis. Recruitment will continue until this number is reached. Assuming an 80% consent rate, we expect to enrol at least 54 participants within 12 months.

Participants in the intervention group will start with an individual pre-assessment with a registered dietitian, focusing on their preferences and values. This aims to build a partnership in care through the participant´s narrative. Next, they will attend an education session on the sustainable, healthy Nordic diet. During this session, the participant will develop an individual health plan together with the dietitian as part of shared decision-making. These handwritten plans will be copied, with one given to the participant and one kept by the dietitian for medical records.

The health plans will be reviewed twice during the study period, allowing for updates with new goals or more realistic targets. These updates will be documented by the dietitian. Participants will receive monthly text message reminders to enhance the intervention's efficacy.

Control group participants will receive short dietary information as part of routine clinical practice. The study duration for all participants is six months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes.
* Diabetes duration for more than 12 months at screening.
* Adults 18 years or older.
* HbA1c more than 57mmol/mol.
* Use of continuous glucose monitoring (CGM) sensor for more than three months at screening and during the study period.
* Use of basal and bolus insulin regimen for more than three months at screening and during the study period.
* Written Informed Consent.

Exclusion Criteria:

* Women of childbearing potential: ongoing pregnancy or planned pregnancy during the study period.
* Cognitive impairment or other disease that study physician find non-compatible with participation.
* Planned change in glucose lowering treatment during study period (change of mealtime insulin analogue with same pharmacodynamic profile allowed).
* Planned change of CGM sensor during the study.
* Food allergies or intolerances that are incompatible with adhering to Nordic nutrition recommendations.
* Current or planned treatment with corticosteroids during the study (other than for replacement therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time in range - Percentage of time spent with blood glucose levels between 3.9-10 mmol/l. | Week 1, 12 and 24.
  Percentage of time spent with glucose levels between 3.9-10 mmol/l measured with continuous glucose monitor (CGM) over 10-14 days.

SECONDARY OUTCOMES:
Adherence to a Nordic diet. | Week 1 and 24.
  Evaluation and analysis of diet data from Food frequency questionnaire (FFQ) and food diary.
Glycosylated Hemoglobin (HbA1c). | Week 1 and 24.
  HbA1c represents overall glycaemic control over the last three months.
Time above range - percentage of time spent with blood glucose levels above 10.0 mmol/L and 13.9 mmol/L respectively. | Week 1, 12 and 24.
  Percentage of time with high blood glucose levels, measured with continuous glucose monitor over 10-14 days.
Time below range - percentage of time spent with blood glucose levels below 3.9 mmol/L and 3.0 mmol/L respectively. | Week 1, 12 and 24.
  Percentage of time with low blood glucose levels, measured with continuous glucose monitor over 10-14 days.
Blood lipids. | Week 1 and 24.
  Blood lipids (total cholesterol, high-density cholesterol, low-density cholesterol, triglycerides, non-HDL cholesterol, cholesterol/HDL ratio) assessed in a clinical laboratory.
Blood pressure. | Week 1 and 24.
  Systolic and diastolic blood pressure measured at hospital clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Stoltz Sjöström, Associate professor, Principal Investigator — Department of Food, Nutrition and Culinary Science, Umeå University, Sweden
Locations (1):
- Hospital of Enköping, Enköping, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No